CLINICAL TRIAL: NCT03383094
Title: Phase II Randomized Trial of Radiotherapy With Concurrent and Adjuvant Pembrolizumab (Keytruda®) Versus Concurrent Chemotherapy in Patients With Advanced/Intermediate-Risk p16+ Head and Neck Squamous Cell Carcinoma (KEYCHAIN)
Brief Title: Chemoradiation vs Immunotherapy and Radiation for Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Loren Mell, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Loren Mell, MD, Director, Division of Clinical and Translational Research/ Department of Radiation Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170862
Record Dates: First submitted 2017-12-18; First posted 2017-12-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Cancer; Cancer of Head and Neck; Cancer, Advanced; Cancer, Metastatic; Tumor; Tumor Recurrence; Tumor Neck; Tumor Metastasis; Oral Cancer; Oropharyngeal Cancer; Oropharynx Cancer; Oropharynx Cancer, Stage III; Oropharynx Cancer, Recurrent; Oropharynx Cancer, Metastatic
Keywords: cancer; Head and Neck; Pembrolizumab; Cisplatin; Radiotherapy; Head and Neck Squamous Cell Carcinoma; p16+; immunotherapy; pd-1; chemotherapy; T1; T2; T3; N2; M0; T4; N3; N1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms; Head and Neck Neoplasms; Neoplasm Metastasis; Recurrence; Mouth Neoplasms; Oropharyngeal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Immunotherapy; Radiotherapy; Cisplatin; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control-radiotherapy/cisplatin (Active Comparator): Intensity-modulated radiation therapy to 70 Gy in 33-35 fractions over 6.5 weeks plus concurrent cisplatin 100 mg/m2 every 3 weeks for 3 cycles (7 weeks)
  Interventions: Radiation: Radiation therapy; Drug: Cisplatin
- Experimental-Radiotherapy/pembrolizumab (Experimental): Intensity-modulated radiation therapy to 70 Gy in 33-35 fractions over 6.5 weeks plus concurrent and adjuvant pembrolizumab 200 mg IV infusion every 3 weeks x 20 cycles
  Interventions: Drug: Pembrolizumab; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV infusion every 3 weeks x 20 cycles
  Other Names: Immunotherapy
  Arms: Experimental-Radiotherapy/pembrolizumab
Radiation: Radiation therapy — 70 Gy in 33-35 fractions
  Other Names: Radiotherapy
Drug: Cisplatin — 100 mg/m2 Weeks 1, 4, and 7.
  Other Names: Chemotherapy
  Arms: Control-radiotherapy/cisplatin

SUMMARY:
The purpose of this study is to compare any good or bad effects of using pembrolizumab (an experimental drug) and radiation therapy (RT), compared to using cisplatin chemotherapy and radiation therapy (RT) in the treatment of patients with head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
This study is a prospective, multi-institutional, open-label, randomized phase II trial that will evaluate the efficacy of concurrent and adjuvant pembrolizumab with radiation therapy (RT) versus RT plus cisplatin in intermediate/high-riskp16-positive locoregionally advanced head and neck squamous cell carcinoma (HNSCC). The primary endpoint is progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* p16-positive squamous cell carcinoma of the pharynx, larynx or oral cavity
* High-Intermediate Risk Disease, defined as:

  * T1-T3 N2 M0 or T3 N1 M0 or any stage III (T4 or N3) p16+ squamous cell carcinoma of the oropharynx (AJCC 8th edition staging system)
  * T1-2 N1-3 M0 or T3-4 N0-3 M0 (stage III-IVB) p16+ squamous cell carcinoma of the hypopharynx or larynx
  * T1-2 N2-3 M0 or T3-4 N0-3 M0 (stage III-IVB) p16+ squamous cell carcinoma of the nasopharynx
  * Inoperable T4 N0-3 M0 (stage IVA-IVB) p16+ squamous cell carcinoma of the oral cavity
* Measurable disease based on RECIST 1.1
* Adequate hematologic function within 28 days prior to registration
* Adequate renal and hepatic function
* Female subject of childbearing potential should have a negative pregnancy test
* Female subjects of childbearing potential must agree to use an adequate method of contraception for the course of the study
* Male subjects must agree to use an adequate method of contraception for the course of the study

Exclusion Criteria:

* Prior malignancy within the past 3 years (except non-melanomatous skin cancer and early stage treated prostate cancer);
* Prior head and neck radiation, chemotherapy, or immunotherapy;
* Prior oncologic (radical) surgery to the primary site;
* Documented evidence of distant metastases;
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
  * Transmural myocardial infarction within the last 6 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration;
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol.
* Any medical or psychiatric illness, which, in the opinion of the principal investigator, would compromise the patient's ability to tolerate this treatment;
* Psychiatric/social situations that would limit compliance with study requirements
* Hypersensitivity to pembrolizumab or any of its excipients.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 3 years
  time from randomization to progression/relapse or death from any cause.

SECONDARY OUTCOMES:
overall survival | 3 years
  time from randomization to death from any cause
Acute toxicity | 3 months
  Toxicities due to therapy occurring within 3 months of therapy completion based on CTCAE criteria using questionnaires
Late toxicity | 3 years
  Toxicity due to therapy occurring greater than 3 months after completion of therapy based on CTCAE criteria using questionnaires
Patterns of failure | 3 years
  Local and regional and distant recurrence of cancer and causes of death from competing events

OTHER OUTCOMES:
PD-L1 expression correlations | 3 years
  compare the outcomes with RT/pembrolizumab in patients with tumors as a function of PD-L1 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Loren Mell, MD, Principal Investigator — University of California, San Diego
Locations (6):
- United States (6):
  - University of Arizona Cancer Center, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - H. Lee Moffitt Cancer Center & Research Facility, Tampa, Florida
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No